CLINICAL TRIAL: NCT05243472
Title: Clinical Efficacy of Protein-Enriched Lacto-Vegetarian Soup on Muscle Mass and Muscle Strength Among Community-Dwelling Older Adults:A 12-Week Randomized Controlled Trial
Brief Title: Impact of Protein-Enriched Lacto-Vegetarian Soup on Muscle Mass and Muscle Strength Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Collaborators: Laurel Corporation, Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB110-246-A
Record Dates: First submitted 2022-01-06; First posted 2022-02-17 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Sarcopenia; Muscle Loss; Malnutrition
Keywords: Older adults; Sarcopenia; Malnutrition
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Malnutrition

STUDY DESIGN:
Intervention Model Description: This program is designed as a parallel randomized intervention. The primary purpose of this program is Prevention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the control group will not receive any intervention during the study period.
- Protein nutritional supplement group (Experimental): Participants in the intervention group will receive protein-enriched soups (24-30g of protein) per day for 12 weeks. Protein may come from either soy, bean or milk products.
  Interventions: Dietary Supplement: Protein nutritional supplement

INTERVENTIONS:
Dietary Supplement: Protein nutritional supplement — Participants in the intervention group will receive protein-enriched soups (24-30g of protein). Protein may come from either soy, bean or milk products.
  Arms: Protein nutritional supplement group

SUMMARY:
The study is a 12-week randomized controlled trial designed to evaluate the clinical effects of protein-enriched Lacto-vegetarian soups on body composition, muscle strength, and physical performance among community-dwelling older adults. Participants are randomly assigned to either an intervention group, which is provided one commercial soup (24-30g of protein) per day for 12 weeks, or the control group, which does not receive this supplement. The investigators also assess the frail status, Mini-Mental Status Examination, Geriatric Depression Scale, Mini Nutritional Assessment, WHOQOL-BREF, and blood tests as outcome measures.

DETAILED DESCRIPTION:
As age increases, the muscle mass of the individual will gradually decrease, which will affect muscle strength and function. If the condition continues to deteriorate, the individual may develop a syndrome of "sarcopenia" in the elderly. In addition to age, risk factors related to sarcopenia include living alone, excessive drinking, lack of physical activity, malnutrition, and oral and dental problems. Among them, lack of physical activity and malnutrition are considered potential risk factors for preventing or improving sarcopenia. Sufficient protein intake is an important method for frail elderly people to improve malnutrition and further prevent or reverse sarcopenia. There were few studies in the past. Some studies had enrolled older adults with sarcopenia, but the participants did not necessarily have nutritional risks; other studies had enrolled individuals with nutritional risks but without complete evaluation for sarcopenia (especially muscle mass). In addition, the components of nutritional supplements should also be adjusted in response to different dietary preferences. For example, past studies have rarely provided protein-enriched nutritional supplements that can be used by Lacto-vegetarian. Therefore, this study aims to evaluate the clinical effects of protein-enriched Lacto-vegetarian soups on body composition, muscle strength, and physical performance among community-dwelling older adults with risk of sarcopenia and malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* People aged 65 years or older
* People with nutritional risk: Mini Nutritional Assessment (MNA) is less than or equal to eleven points.
* People with risk of sarcopenia: SARC-F questionnaire greater than or equal to four points or SARC-CalF questionnaire greater than or equal to eleven points.
* People can understand the research process, meet the requirements of the research, and can sign the informed consent and participate in the following tracking.

Exclusion Criteria:

* People that are unable to cooperate with or accept lacto-vegetarian-based/nuts/gluten foods, such as those who are allergic to dietary content, nuts or gluten, etc.
* According to the PI's judgment, people with severe or poorly controlled conditions include acute diseases, severe infections, severe abnormal laboratory tests, or serious medical conditions with the following systems: cardiovascular, pulmonary, hepatic, nervous, mental, metabolic, renal, musculoskeletal, gastrointestinal, etc.
* People with liver cirrhosis
* People with chronic kidney diseases (eGFR <30ml/min/1.73m2)
* People with severe visual or hearing impairment that prevent the completion of assessment and testing
* People with malignant tumors that have just been diagnosed or are undergoing treatment or are still at risk of recurrence
* People are known to be infected with human immunodeficiency virus or HIV antibody-positive.
* People have received hormone therapy within three months before the trial or are expected to receive hormone therapy during the trial
* People are currently or expected to join any other physical training courses or nutrition plans during the trial
* Others are based on the judgment of the PI that participating in this trial may adversely affect the safety of the subjects, hinder the progress of the experiment, or interfere with the evaluation of the outcomes of the trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline muscle strength measure by hand grip strength after 12 weeks | baseline, 12 weeks
  measured by hand grip strength
Change from baseline walking speed after 12 weeks | baseline, 12 weeks
  measured by six-meter walking speed
Changes from baseline physical performance after 12 weeks | baseline, 12 weeks
  measured by Short Physical Performance Battery
Changes from baseline frailty after 12 weeks | baseline, 12 weeks
  measured by Clinical Frailty Scale
Changes from baseline frail status after 12 weeks | baseline, 12 weeks
  measured by Fatigue, Resistance, Ambulation, Illnesses, & Loss of Weight scale
Changes from baseline cognition after 12 weeks | baseline, 12 weeks
  measured by Mini-Mental Status Examination
Changes from baseline depression after 12 weeks | baseline, 12 weeks
  measured by Geriatric Depression Scale
Changes from baseline quality of life after 12 weeks | baseline, 12 weeks
  measured by WHOQOL-BREF (Taiwan Version)
Changes from baseline physical activity after 12 weeks | baseline, 12 weeks
  measured by the International Physical Activity Questionnaire (IPAQ)
Changes from baseline nutritional status after 12 weeks | baseline, 12 weeks
  measured by Mini-Nutritional Assessment-Short Form (MNA-SF)
Changes from baseline dietary assessment after 12 weeks | baseline, 12 weeks
  measured by Food Frequency Questionnaires (FFQ)

SECONDARY OUTCOMES:
Change from baseline complete blood count 12 weeks | baseline, 12 weeks
  Change from baseline complete blood count 12 weeks
Change from baseline differential count 12 weeks | baseline, 12 weeks
  Change from baseline differential count 12 weeks
Change from baseline percentage of glycated hemoglobin (HbA1c) after 12 weeks | baseline, 12 weeks
  Change from baseline percentage of glycated hemoglobin (HbA1c) after 12 weeks
Change from baseline concentration of alanine aminotransferase (ALT) after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of alanine aminotransferase (ALT) after 12 weeks
Change from baseline concentration of aspartate aminotransferase (AST) after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of aspartate aminotransferase (AST) after 12 weeks
Change from baseline concentration of blood urea nitrogen (BUN) after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of blood urea nitrogen (BUN) after 12 weeks
Change from baseline concentration of Creatinine after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of Creatinine after 12 weeks
Change from baseline concentration of sodium after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of sodium after 12 weeks
Change from baseline concentration of potassium after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of potassium after 12 weeks
Change from baseline concentration of uric acid after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of uric acid after 12 weeks
Change from baseline concentration of total protein after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of total protein after 12 weeks
Change from baseline concentration of albumin after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of albumin after 12 weeks
Change from baseline concentration of globulin after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of globulin after 12 weeks
Change from baseline concentration of cholesterol after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of cholesterol after 12 weeks
Change from baseline concentration of high-density lipoprotein cholesterol (HDL-C) after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of high-density lipoprotein cholesterol (HDL-C) after 12 weeks
Change from baseline concentration of low-density lipoprotein cholesterol (LDL-C) after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of low-density lipoprotein cholesterol (LDL-C) after 12 weeks
Change from baseline concentration of triglyceride after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of triglyceride after 12 weeks
Change from baseline concentration of fasting glucose after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of fasting glucose after 12 weeks
Change from baseline concentration of high-sensitivity C-reactive protein (hs-CRP) after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of high-sensitivity C-reactive protein (hs-CRP) after 12 weeks
Change from baseline concentration of fasting insulin after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of fasting insulin after 12 weeks
Change from baseline concentration of Vitamin D after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of Vitamin D after 12 weeks
Change from baseline concentration of Vitamin B12 after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of Vitamin B12 after 12 weeks
Change from baseline concentration of homocysteine after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of homocysteine after 12 weeks
Change from baseline concentration of cystatin C after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of cystatin C after 12 weeks
Change from baseline concentration of DHEA-S after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of DHEA-S after 12 weeks
Change from baseline body weight after 12 weeks | baseline, 12 weeks
  Change from baseline body weight after 12 weeks
Change from baseline fat mass after 12 weeks | baseline, 12 weeks
  Change from baseline fat mass after 12 weeks
Change from baseline muscle mass after 12 weeks | baseline, 12 weeks
  Change from baseline muscle mass after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hui Loh, MD.PhD., Principal Investigator — Buddhist Tzu Chi General Hospital
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No